CLINICAL TRIAL: NCT06618846
Title: Impact of Bariatric and Metabolic Surgery on the Reduction of Premature Aging.
Status: Completed | Type: Observational
Sponsor: University Hospital in Krakow (Other)
Collaborators: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Alicja Dudek, Principal Investigator, PhD Candidate, Medical Doctor, University Hospital in Krakow
Other Study IDs: DI2018 013048
Record Dates: First submitted 2024-09-20; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: biological age markers; bariatric surgery; metabolic surgery; premature aging
MeSH Terms: conditions — Obesity; Aging, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples to determine telomere lenght RNA samples to determine microRNA from telomerase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- bariatric patients: Patients who were qualified for bariatric or metabolic surgery
  Interventions: Procedure: laparoscopic sleeve gastric bypass

INTERVENTIONS:
Procedure: laparoscopic sleeve gastric bypass — This is the observational study that investigate the impact of laparoscopic Sleeve Gastrectomy (LSG) or laparoscopic Roux-en-Y Gastric Bypass on premature aging by the assesment of biological age markers (telomere lenght, IL-6, TNFalpha, total oxidative status, DNA damage, cognitive function)

SUMMARY:
We invite the participants to take a part in a research study conducted at the 2nd Department of General Surgery of the Jagiellonian University Medical College. This study is for patients who are scheduled for laparoscopic sleeve gastrectomy (LSG) or laparoscopic Roux-en-Y gastric bypass (LRYGB) to treat morbid obesity.

Study Purpose:

The study aims to assess how obesity surgery impacts aging, specifically by examining changes in telomere length (a marker of molecular age). The research will also evaluate other aspects of ageing, such as metabolic, psychological, and biochemical factors, to understand how surgery may reverse aging.

Study Design:

The study will be observational and consist of two phases. In the first phase (pre-surgery), clinical and metabolic data will be collected, including blood samples for inflammatory markers, DNA damage tests, and gene expression analysis. Psychological and metabolic age will also be assessed.

The second phase will take place 24 months after surgery, with similar tests repeated.

A third stage will focus on a detailed gene expression analysis for the 12 patients showing the most significant changes in telomere length and DNA damage.

What Will Be The Participants Asked For:

The participants will be asked to provide blood samples (for the analysis of: inflammatory markers: C-reactive protein, Tumor necrosis factor alpha, Interleukin-6, marker of DNA damage and total oxidative capacity; the other 2 probes will be collected to analyze telomere length and the probe for RNA to identify gene expression connected to telomere elongation), as well as to complete psychological and metabolic assessments (body composition analysis) in two time points - before and 24 months after surgery. Tests and assessments will take approximately 30 minutes.

Voluntary Participation:

Participation is entirely voluntary. The participation will NOT affect the treatment at any timepoints.

This study seeks to provide new insights into premature aging in patients with morbid obesity, which could help improve care for future bariatric patients. The participants might gain more knowledge about the outcomes of their surgical treatment.

DETAILED DESCRIPTION:
We would like to invite the participants to take part in a research study carried out at the 2nd Department of General Surgery of the Jagiellonian University CM.

Participation in the study is offered to patients who have qualified for surgical treatment of morbid obesity and have been accepted for laparoscopic sleeve gastrectomy (LSG) or laparoscopic Roux-en-Y gastric bypass (LRYGB) in the Department of Endoscopic, Metabolic and Soft Tissue Surgery. It is well known that morbid obesity contributes to premature aging. One of the topics addressed in recent scientific research is the mechanism of reversal of the aging process in patients undergoing LSG or LRYGB surgery. Assessments of the progression of aging can be carried out by evaluating the age of the body in different contexts. For this purpose, metabolic age - indicating the level of basal metabolism, psychological age - the ability to cognitively function, focus attention, remember, biochemical age - the level of oxidative stress on cells - are determined. A much better parameter for assessing organismal age is telomere length (TL) - molecular age. Telomeres are specialised structures located at the ends of chromosomes - the intracellular structures that carry genetic information. Telomere shortening with age is part of the normal aging process. It has been shown that patients suffering from morbid obesity have shorter telomere lengths compared to people of the same age who have never suffered from obesity, and that telomeres might lengthen after bariatric surgery. However, it is unclear what is responsible for the effect of telomere lengthening, thereby reversing the aging process. The proposed study aims to assess the effect of metabolic surgery on telomere length change and other markers of aging (metabolic age, psychological age, biochemical age, molecular age). The secondary objectives of the study will be to understand the mechanisms responsible for reversing the aging process in bariatric and metabolic surgery patients.

An observational study consisting of two phases was planned. In the first stage, baseline anthropometric and clinical data will be collected on the day of admission to the surgical ward, including the following parameters: age, sex, body weight, height, BMI, duration of obesity, family history of obesity, preoperative weight loss, information on concomitant diseases and medications taken. For the assessment of biochemical and molecular aging, the participants will be asked to consent to the collection of three tubes of peripheral blood.

One blood sample will be preserved in serum tubes for the analysis of inflammatory parameters such as Interleukin-6 (IL-6), C-reactive protein (CRP), Tumor necrosis factor alpha (TNFalpha) and for the determination of the blood antioxidant capacity - total oxidative status (TOS). A second blood sample will be collected into tubes containing an anticoagulant in the form of EDTA for the isolation of DNA for the assessment of DNA damage marker and telomere length. A third blood sample will be preserved in special RNA Pax tubes for testing of expression of genes related to telomere lenghtening. The other markers of aging will include: metabolic age (assessed by bioimpedance scanning, TANITA) and the psychological age determined by using special psychological tests (CTT Colour Connectivity Test and Winscosin Card Sorting Test) for the assessment of cognitive function. Ale the tests will take approximately 30 minutes to be completed.

The second stage of the study will take place 24 months after the operation at the follow-up visit, when all the steps described above will be performed again.

After receiving the results from the first two stages of the study, the third stage will identify the twelve patients (six LSG patients and six LRYGB patients) who will show the greatest difference in telomere length 24 months after surgery and the greatest change in the degree of DNA damage. An in-depth analysis of the expression of genes responsible for telomere lengthening will be carried out in these patients.

This study is an attempt to identify new clinical aspects of the surgical treatment undertaken.The results obtained are expected to help understand the mechanism of premature aging in people suffering from higher stages of obesity, which may in future contribute to the individualisation of perioperative care for bariatric patients and the introduction of prevention programmes.

The decision to participate in the study is completely voluntary. Everyone assesses for themselves whether they have understood the doctor's explanations and the written information provided about the trial. The course of treatment is not altered if a decision is made not to participate.

ELIGIBILITY:
Inclusion Criteria:

* BMI values > 40 kg m2 or BMI > 35 kg/m2 with obesity related complications, age range between 18 and 60
* consent to participant in the study

Exclusion Criteria:

* reversal bariatric surgery or previous bariatric surgery, pregnancy during follow up period, uncontrolled thyroid disorders, kidney diseases, pancreatitis, cancer, depression, neurological disorders, any condition affecting cognitive function or consumed medications impairing cognitive functioning
* lack of consent to participant in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients aged between 18-65 years old who were qualified for the bariatric or metabolic surgery with criteria (BMI values > 40 kg m2 or BMI > 35 kg/m2 with obesity related complication), who met the inclusion criteria at the follow up visit after 2 years. All study participants participated in an aftercare programme, which included meetings with a dietician and a psychologist.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-11-17 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
The impact of bariatric and metabolic surgery on reduction of premature aging | Two years
  The primary outcome will be to determine the effect of metabolic surgery after two years on: telomere length in base pairs, DNA damage in picogram, Interleukin-6 in picogram per mililitr, C-reactive protein in miligram per deciliter, tumor necrosis factor alpha in picogram per milliliter, total oxidative status in micromole per liter and the results of Color Trial Test presented as seconds of test completion and achieved centile.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Krakow, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided